CLINICAL TRIAL: NCT06946654
Title: Geriatric Assessment (GA) for Elderly Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation: a Prospective Study.
Brief Title: Geriatric Assessment (GA) for Elderly Patients Undergoing Allo-HSCT
Acronym: GA
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Yuqian, Associate Professor, Peking University People's Hospital
Other Study IDs: 2025PHB131-001
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Elderly; Geriatric Assessment; ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION
Keywords: elderly; Geriatric Assessment; allo-HSCT
MeSH Terms: interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric Assessment
  Interventions: Procedure: Geriatric Assessment

INTERVENTIONS:
Procedure: Geriatric Assessment — This is a study held in all patients undergoing allogenic hematopoietic stem cell transplantation. Pre-transplant assessment: (1)Patients-related assessment: (a) Age; (b) Functional status (BADL score; IADL score; KPS score; ECOG PS score); (c) Comorbidities (HCT-CI score); (d) Nutritional Status (Body weight; BMI; NRS-2002; MNA-SF; MUST); (e) Psychological Status (SF36-MCS; GDS; PHQ-9; GAD-7); (f) Cognitive Function (MMSE; BMOC); (g) Social Support Level (MOS-SSS; MSPSS); (h) Total Number of Medications Used. (2) Disease-Related Factors Assessment: Primary Disease Diagnosis; ELN Risk Stratification (assessed only for AML patients); Disease Status. (3) Donor-Related Factors Assessment: Donor Age; Donor Sex; Donor-Recipient Blood Type Compatibility; Donor Type; DSA. (4) Treatment-Related Factors Assessment: Conditioning Regimen; GVHD Prophylaxis Regimen; Graft Type.

SUMMARY:
This comprehensive, multidimensional evaluation assesses patient-related factors, disease-related factors, donor-related factors, and treatment-related factors. The study aims to identify potential risk factors influencing transplant outcomes in elderly patients and enhance the outcomes of allo-HSCT.

DETAILED DESCRIPTION:
This comprehensive, multidimensional evaluation assesses patient-related factors (e.g., age, physical function, and comorbidity index), disease-related factors (e.g., primary diagnosis and blast count), donor-related factors (e.g., donor age, sex, ABO, and type), and treatment-related factors (e.g., conditioning regimen, graft source, and GVHD prophylaxis). The study aims to identify potential risk factors influencing transplant outcomes in elderly patients, establish a comprehensive geriatric assessment model, and guide personalized pre-transplant treatment strategies to reduce transplant-related mortality (TRM). Ultimately, we hope this study could help enhance the outcomes of allogenic hematopoietic stem cell transplantation (allo-HSCT).

ELIGIBILITY:
Inclusion Criteria:

* (a)Age ≥55 years.
* (b)Hematologic disorders with established indications for transplantation, including malignant and non-malignant hematologic diseases. (c)Willingness to provide informed consent.

Exclusion Criteria: (a)Pregnancy. (b) Uncontrolled active infection. (c) Lack of informed consent. (d)Deemed ineligible for transplantation after investigator assessment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients with hematologic disorders with established indications for transplantation, including malignant and non-malignant hematologic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Transplant-related mortality | From HSCT to the follow-up assessment at 12 months post-treatment.
  Transplant-related mortality (TRM) is defined as death due to any transplantation-related cause other than disease relapse. Transplant-related mortality will be calculated using a competing risks model.

SECONDARY OUTCOMES:
Engraftment | From HSCT to the follow-up assessment at 12 months post-treatment.
  Platelet engraftment was defined as the first of seven consecutive days with a platelet count >20 × 109/L without transfusion support. Neutrophil engraftment was defined as the first of three consecutive days with an ANC > 0.5 × 109/L.
GVHD | From HSCT to the follow-up assessment at 12 months post-treatment.
  Acute GVHD was classified as symptom presentation before 100 days after haplo-HSCT and chronic GVHD was classified as symptom presentation >100 days after haplo-HSCT. Each organ (skin, liver, and gut) was staged 1 through 4 for Acute GVHD according to modified criteria based on the schema of the Mount Sinai Acute GVHD International Consortium (MAGIC), and patients were also assigned a grade of acute GVHD (I through IV) based on overall severity. Chronic GVHD was graded in accordance with the National Institutes of Health (NIH) Chronic Graft-versus-Host Disease Consensus Criteria.
Overall Survival | From HSCT to the follow-up assessment at 12 months post-treatment.
  The time from haplo-HSCT to death from any cause in patients with AML. Overall survival will be calculated using the Kaplan-Meier method.
Cumulative Incidence of Relapse | From HSCT to the follow-up assessment at 12 months post-treatment.
  Relapse was defined as disease recurrence.
Disease-Free Survival | From HSCT to the follow-up assessment at 12 months post-treatment.
  Disease-free survival (DFS) was defined as the time from transplantation to relapse, disease progression, or death, whichever occurred first.
Viral Infection | From HSCT to the follow-up assessment at 12 months post-treatment.
  Detection of CMV-DNA and EBV-DNA in peripheral blood twice a week.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China